CLINICAL TRIAL: NCT02345551
Title: The Feasibility of a Telephone and Web-based Physical Activity Intervention for Female Shift Workers.
Brief Title: A Physical Activity Intervention for Female Shift Workers
Acronym: SWPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H14-03408
Record Dates: First submitted 2014-12-16; First posted 2015-01-26 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Physical Activity
Keywords: Exercise; Sleep; Telemedicine; Behavior; Shift work
MeSH Terms: conditions — Motor Activity; Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): The behaviour change intervention to promote an increase in moderate-vigorous physical activity (to meet the cancer prevention guidelines of 150 min/week) will be guided by the Health Action Process Approach (HAPA) model. This model aims to promote behaviour change through increasing self-efficacy for intention, planning and maintenance of physical activity. As a compliment to the behavioural counseling sessions, participants will be asked to track their physical activity using the FitBit, a wrist-worn activity monitor (www.fitbit.com) which monitors step counts, distance covered, and active minutes and also tracks sleep. The FitBit synchronizes wirelessly to the participants' computer and/or smartphones, thus minimizing the need for daily data entry tracking by participants.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate-vigorous aerobic activity in line with published guidelines for cancer prevention

SUMMARY:
This project will assess the feasibility of a 12-week physical activity program developed specifically for females exposed to a known occupational carcinogen - shiftwork. Physical activity has been shown to decrease cancer risk, but the investigators research has found that female shift workers face unique barriers to participating in physical activity. This project will use a combination of telephone-based behavioural counseling sessions with a physical activity coach, and innovative web-based physical activity tracking software using a Fitbit and website or smartphone app to address commonly reported barriers to physical activity in female shift workers.

DETAILED DESCRIPTION:
Currently 4.1 million Canadians are employed in shiftwork. Shiftwork, defined as the organization of working time to cover more than the usual 8-hour workday and up to a 24-hour period, is prevalent in health care, emergency services, manufacturing, retail and hospitality. Given the growing demand for goods and services at all hours in today's society, the number of shift workers is unlikely to decrease. There is emerging evidence that shiftwork has many negative health implications, including a higher risk of cancer and other chronic diseases. A recent systematic review by members of the investigators study team reported preliminary evidence that changes in shift scheduling, timed exposure to bright light during a night shift, and pharmacological therapy for sleep, help to improve sleep and markers of circadian rhythm dysfunction in shift workers. However changes in shift schedules, and exposure to bright light may be difficult to implement in certain workplaces (i.e., specific hospital environments, police patrol cars) and long-term effects of pharmacological therapy are unknown. To date there is very limited research on effective health promotion strategies in this occupational group, who face unique challenges to engaging in health behaviour change. There is an urgent need to develop and evaluate interventions to improve health and reduce cancer risk in this high-risk population. Participation in regular physical activity is known to decrease risk of cancer and other chronic diseases, and may be a simple and cost-effective intervention that could be implemented in workplaces and by individual workers to mitigate this increased risk. Shift workers have unique barriers to participating in physical activity; therefore the feasibility of implementing such interventions must first be investigated.

Objective 1: To assess the feasibility of a 12-week telephone and web-based physical activity intervention in female shift workers, including recruitment, retention, adherence and acceptability of the intervention.

Objective 2: To explore changes in physical activity (min/week), health behaviours (i.e., sedentary time, sleep), and quality of life that may occur during the intervention in preparation for a full randomized controlled trial (RCT) if the intervention is found to be feasible.

Research Methods:

As the aim of the study is to evaluate feasibility, the investigators will use a single-group pre-post intervention design.

The behaviour change intervention to promote an increase in min/week of moderate-vigorous physical activity will be guided by the Health Action Process Approach (HAPA) model. This model aims to promote behaviour change through increasing self-efficacy for intention, planning and maintenance of physical activity. The goal is for participants to meet Canada's Physical Activity Guidelines for adults of 150 min/week of moderate-vigorous physical activity.

As a compliment to the behavioural counseling sessions, participants will be asked to track their physical activity. All participants will be given a FitBit wrist-worn activity monitor (www.fitbit.com) which monitors step counts, distance covered, and active minutes and also tracks sleep. The FitBit synchronizes wirelessly to the participants' computer and/or smartphones, thus minimizing the need for daily data entry tracking by participants.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Live/work in the greater Vancouver area or willing to come to Vancouver for baseline visit
* Able to read, speak and understand english
* Work a job requiring high circadian disruption (at least 5 night shifts per month) for at least 3 years
* Telephone and internet access

Exclusion Criteria:

* >90 minutes per week of moderate-vigorous physical activity
* Answer 'Yes' to any question on the PAR-Q
* Pregnant or planning to become pregnant
* BMI > 40.0 kg/m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Feasibility: A composite outcome of overall feasibility will be assessed as the primary outcome. | Baseline, 12 weeks
  We will consider the intervention to be feasible if all of the following conditions are met: 1) Achieve a recruitment goal of 20 participants in three months; 2) Achieve a retention rate of 80% of enrolled participants; 3) Achieve > 80% adherence to behavioral counseling sessions; and 4) >80% of participants rank their satisfaction with the study as "Satisfied" (4) or "Very Satisfied" (5) on a five-point Likert scale.

SECONDARY OUTCOMES:
Physical Activity (MET hours per week) | Baseline, 12 weeks
  Accelerometry (Actigraph GT3x+)
Sedentary Time | Baseline, 12 weeks
  Accelerometry (Actigraph GT3x+)
Sleep quantity and quality | Baseline, 12 weeks
  Pittsburgh sleep quality index
Quality of Life | Baseline, 12 weeks
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Campbell, BScPT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Clinical Exercise Physiology Lab, Vancouver, British Columbia, Canada